CLINICAL TRIAL: NCT00584831
Title: Development and Implementation of a Clinical Test to Investigate the Change in Vision With Soft Toric Contact Lenses During Eye Movements
Brief Title: Effect of Eye Movement on Toric Lens Orientation and Visual Acuity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0725; J07-416
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2011-11-01 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Astigmatism
Keywords: astigmatism; visual acuity; orientation; contact lenses
MeSH Terms: conditions — Astigmatism; Orientation, Spatial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (19):
- Group 2 LSBO (Active Comparator): contact lenses worn in this order: lotrafilcon B toric, senofilcon A toric, balafilcon A toric, omafilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 3 LOSB (Active Comparator): contact lenses worn in this order: lotrafilcon B toric, omafilcon A toric, senofilcon A toric, balafilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 4 LBSO (Active Comparator): contact lenses worn in this order: lotrafilcon B toric, balafilcon A toric, senofilcon A toric, omafilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 5 LBOS (Active Comparator): contact lenses worn in this order: lotrafilcon B toric, balafilcon A toric, omafilcon A toric, senofilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 6 SLOB (Active Comparator): contact lenses worn in this order: senofilcon A toric, lotrafilcon B toric, omafilcon A toric, balafilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 7 SLBO (Active Comparator): contact lenses worn in this order: senofilcon A toric, lotrafilcon B toric, balafilcon A toric, omafilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 8 SOLB (Active Comparator): contact lenses worn in this order: senofilcon A toric, omafilcon A toric, lotrafilcon B toric, balafilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 9 SBLO (Active Comparator): contact lenses worn in this order: senofilcon A toric, balafilcon A toric, lotrafilcon B toric, omafilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 10 SBOL (Active Comparator): contact lenses worn in this order: senofilcon A toric, balafilcon A toric, omafilcon A toric, lotrafilcon B toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 11 OSLB (Active Comparator): contact lenses worn in this order: omafilcon A toric, senofilcon A toric, lotrafilcon B toric, balafilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 12 OSBL (Active Comparator): contact lenses worn in this order: omafilcon A toric, senofilcon A toric, balafilcon A toric, lotrafilcon B toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 13 OBLS (Active Comparator): contact lenses worn in this order: omafilcon A toric, balafilcon A toric, lotrafilcon B toric, senofilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 14 OBSL (Active Comparator): contact lenses worn in this order: omafilcon A toric, balafilcon A toric, senofilcon A toric, lotrafilcon B toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 15 BLSO (Active Comparator): contact lenses worn in this order: balafilcon A toric, lotrafilcon B toric, senofilcon A toric, omafilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 16 BLOS (Active Comparator): contact lenses worn in this order: balafilcon A toric, lotrafilcon B toric, omafilcon A toric, senofilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 17 BSOL (Active Comparator): contact lenses worn in this order: balafilcon A toric, senofilcon A toric, omafilcon A toric, lotrafilcon B toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 18 BOLS (Active Comparator): contact lenses worn in this order: balafilcon A toric, omafilcon A toric, lotrafilcon B toric, senofilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 19 BOSL (Active Comparator): contact lenses worn in this order: balafilcon A toric, omafilcon A toric, senofilcon A toric, lotrafilcon B toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B
- Group 1 LSOB (Active Comparator): contact lenses worn in this order: lotrafilcon B toric/senofilcon A toric/omafilconA toric/balafilcon A toric
  Interventions: Device: senofilcon A; Device: balafilcon A; Device: omafilcon A; Device: lotrafilcon B

INTERVENTIONS:
Device: senofilcon A — toric contact lens
Device: balafilcon A — toric contact lens
Device: omafilcon A — toric contact lens
Device: lotrafilcon B — toric contact lens

SUMMARY:
The relative performance of a new toric soft contact lens against toric contact lenses currently available in market, specifically for visual acuity and lens orientation. The study will be conducted in a staged approach (2 stages).

DETAILED DESCRIPTION:
Non-dispensing, single-masked (subject-masked), randomised, controlled study. Two visits.

ELIGIBILITY:
Inclusion Criteria:

1. They are aged between 18-39 years.
2. They understand their rights as a research subject and are willing to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They can attain at least 6/9 in each eye with their spectacle refraction.
5. They have successfully worn contact lenses within six months of starting the study.
6. They can be fitted with toric soft contact lenses to match the available power range.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
7. They are pregnant or lactating.
8. They have grade 2 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
9. They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD MCOptom, Principal Investigator — Eurolens Research, The University of Manchester Dpt. of Optometry and Neuroscience
Locations (1):
- Eurolens Research, The University of Manchester Dpt. of Optometry & Neuroscience, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Group1 LSOB: lotrafilcon b toric, senofilcon A toric, omafilcon A toric, balafilcon A toric
- Group 2 LSBO: lotrafilcon B toric, senofilcon A toric, balafilcon A toric, omafilcon A toric
- Group 4 LBSO: lotrafilcon B toric, balafilcon A toric, senofilcon A toric, omafilcon A toric
- Group 5 LBOS: lotrafilcon B toric, balafilcon A toric, omafilcon A toric, senofilcon A
- Group 7 SLBO: senofilcon A toric, lotrafilcon B toric, balafilcon A toric, omafilcon A toric
- Group 8 SOLB: senofilcon A toric, omafilcon A toric, lotrafilcon B toric, balafilcon A toric
- Group 9 SBLO: senofilcon A toric, balafilcon A toric, lotrafilcon B toric, omafilcon A toric
- Group 10 SBOL: senofilcon A toric, balafilcon A toric, omafilcon A toric, lotrafilcon B toric
- Group 11 OSLB: omafilcon A toric, senofilcon A toric, lotrafilcon B toric, balafilcon A toric
- Group 12 OSBL: omafilcon A toric, senofilcon A toric, balafilcon A toric, lotrafilcon B toric
- Group 13 OBLS: omafilcon A toric, balafilcon A toric, lotrafilcon B toric, senofilcon A toric
- Group 14 OBSL: omafilcon A toric, balafilcon A toric, senofilcon A toric, lotrafilcon B toric
- Group 15 BLSO: balafilcon A toric, lotrafilcon B toric, senofilcon A toric, omafilcon A toric
- Group 16 BLOS: balafilcon A toric, lotrafilcon B toric, omafilcon A toric, senofilcon A toric
- Group 18 BOLS: balafilcon A toric, omafilcon A toric, lotrafilcon B toric, senofilcon A toric
- Group 19 BOSL: balafilcon A toric, omafilcon A toric, senofilcon A toric, lotrafilcon B toric
- Group 3 LOSB: lotrafilcon B toric, omafilcon A toric, senofilcon A toric, balafilcon A toric
- Group 6 SLOB: senofilcon A toric, lotrafilcon b toric, omafilcon A toric, balafilcon A toric
- Group 17 BSOL: balafilcon A toric, senofilcon A toric,omafilcon A toric, lotrafilcon b toric
Period: Intervention 1
Arm/Group | Group1 LSOB | Group 2 LSBO | Group 4 LBSO | Group 5 LBOS | Group 7 SLBO | Group 8 SOLB | Group 9 SBLO | Group 10 SBOL | Group 11 OSLB | Group 12 OSBL | Group 13 OBLS | Group 14 OBSL | Group 15 BLSO | Group 16 BLOS | Group 18 BOLS | Group 19 BOSL | Group 3 LOSB | Group 6 SLOB | Group 17 BSOL
Started | 1 | 3 | 2 | 1 | 2 | 1 | 6 | 2 | 4 | 2 | 2 | 1 | 2 | 1 | 3 | 1 | 4 | 1 | 1
Completed | 1 | 3 | 2 | 1 | 2 | 1 | 6 | 2 | 4 | 2 | 2 | 1 | 2 | 1 | 3 | 1 | 4 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 2
Arm/Group | Group1 LSOB | Group 2 LSBO | Group 4 LBSO | Group 5 LBOS | Group 7 SLBO | Group 8 SOLB | Group 9 SBLO | Group 10 SBOL | Group 11 OSLB | Group 12 OSBL | Group 13 OBLS | Group 14 OBSL | Group 15 BLSO | Group 16 BLOS | Group 18 BOLS | Group 19 BOSL | Group 3 LOSB | Group 6 SLOB | Group 17 BSOL
Started | 1 | 3 | 2 | 1 | 2 | 1 | 6 | 2 | 4 | 2 | 2 | 1 | 2 | 1 | 3 | 1 | 4 | 1 | 1
Completed | 1 | 3 | 2 | 1 | 2 | 1 | 6 | 2 | 4 | 2 | 2 | 1 | 2 | 1 | 3 | 1 | 4 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 3
Arm/Group | Group1 LSOB | Group 2 LSBO | Group 4 LBSO | Group 5 LBOS | Group 7 SLBO | Group 8 SOLB | Group 9 SBLO | Group 10 SBOL | Group 11 OSLB | Group 12 OSBL | Group 13 OBLS | Group 14 OBSL | Group 15 BLSO | Group 16 BLOS | Group 18 BOLS | Group 19 BOSL | Group 3 LOSB | Group 6 SLOB | Group 17 BSOL
Started | 1 | 3 | 2 | 1 | 2 | 1 | 6 | 2 | 4 | 2 | 2 | 1 | 2 | 1 | 3 | 1 | 4 | 1 | 1
Completed | 1 | 3 | 2 | 1 | 2 | 1 | 6 | 2 | 4 | 2 | 2 | 1 | 2 | 1 | 3 | 1 | 4 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 4
Arm/Group | Group1 LSOB | Group 2 LSBO | Group 4 LBSO | Group 5 LBOS | Group 7 SLBO | Group 8 SOLB | Group 9 SBLO | Group 10 SBOL | Group 11 OSLB | Group 12 OSBL | Group 13 OBLS | Group 14 OBSL | Group 15 BLSO | Group 16 BLOS | Group 18 BOLS | Group 19 BOSL | Group 3 LOSB | Group 6 SLOB | Group 17 BSOL
Started | 1 | 3 | 2 | 1 | 2 | 1 | 6 | 2 | 3 | 2 | 2 | 1 | 2 | 1 | 2 | 1 | 4 | 1 | 1
Completed | 1 | 3 | 2 | 1 | 2 | 1 | 6 | 2 | 3 | 2 | 2 | 1 | 2 | 1 | 2 | 1 | 4 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Study Population
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 40

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity After Infero-temporal Version Movement.
Description: logarithm of the minimum angle of resolution (logMar) ideal is 0.0 and represents 20/20 Snellen acuity. logMar values > 0.00 indicate vision poorer than the ideal and values <0.00 indicate vision greater than the ideal.
Time Frame: 10 minutes after insertion
Measure: Mean (Standard Deviation); unit: LogMAR units
Groups:
- Lotrafilcon B: lotrafilcon b toric
- Senofilcon A: senofilcon A toric
- Omafilcon A: omafilcon A toric
- Balafilcon A: balafilcon A toric
Arm/Group | Lotrafilcon B | Senofilcon A | Omafilcon A | Balafilcon A
Number analyzed (Participants) | 35 | 35 | 35 | 35
LogMAR units | 0.12 (0.16) | 0.1 (0.15) | 0.16 (0.17) | 0.14 (0.19)
Statistical Analysis 1: Comparison: Lotrafilcon B vs Senofilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = 0.03, Standard Deviation 0.16
Statistical Analysis 2: Comparison: Lotrafilcon B vs Omafilcon A; Hyposthesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.04, Standard Deviation 0.18
Statistical Analysis 3: Comparison: Lotrafilcon B vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.02, Standard Deviation 0.20
Statistical Analysis 4: Comparison: Senofilcon A vs Omafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.06, Standard Deviation 0.17
Statistical Analysis 5: Comparison: Senofilcon A vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.04, Standard Deviation 0.18
Statistical Analysis 6: Comparison: Omafilcon A vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = 0.02, Standard Deviation 0.18

2. Primary Outcome: Visual Acuity After Infero-nasal Version Movement.
Description: as for outcome 1
Time Frame: 10 minutes after lens insertion
Measure: Mean (Standard Deviation); unit: LogMAR units
Arm/Group | Lotrafilcon B | Senofilcon A | Omafilcon A | Balafilcon A
Number analyzed (Participants) | 35 | 35 | 35 | 35
LogMAR units | 0.12 (0.16) | 0.11 (0.16) | 0.14 (0.17) | 0.15 (0.20)
Statistical Analysis 1: Comparison: Lotrafilcon B vs Senofilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = 0.02, Standard Deviation 0.16
Statistical Analysis 2: Comparison: Lotrafilcon B vs Omafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.01, Standard Deviation 0.17
Statistical Analysis 3: Comparison: Lotrafilcon B vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.03, Standard Deviation 0.17
Statistical Analysis 4: Comparison: Senofilcon A vs Omafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.03, Standard Deviation 0.19
Statistical Analysis 5: Comparison: Senofilcon A vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.04, Standard Deviation 0.20
Statistical Analysis 6: Comparison: Omafilcon A vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.02, Standard Deviation 0.17

3. Primary Outcome: Visual Acuity After Superior-temporal Version Movement
Description: as for outcome 1
Time Frame: 10 minutes after lens insertion
Measure: Mean (Standard Deviation); unit: LogMAR units
Arm/Group | Lotrafilcon B | Senofilcon A | Omafilcon A | Balafilcon A
Number analyzed (Participants) | 35 | 35 | 35 | 35
LogMAR units | 0.11 (0.15) | 0.08 (0.14) | 0.13 (0.17) | 0.14 (0.20)
Statistical Analysis 1: Comparison: Lotrafilcon B vs Senofilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = 0.03, Standard Deviation 0.13
Statistical Analysis 2: Comparison: Lotrafilcon B vs Omafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.01, Standard Deviation 0.15
Statistical Analysis 3: Comparison: Lotrafilcon B vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.02, Standard Deviation 0.17
Statistical Analysis 4: Comparison: Senofilcon A vs Omafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.04, Standard Deviation 0.15
Statistical Analysis 5: Comparison: Senofilcon A vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.06, Standard Deviation 0.17
Statistical Analysis 6: Comparison: Omafilcon A vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.01, Standard Deviation 0.18

4. Primary Outcome: Visual Acuity After Superior-nasal Version Movement.
Description: as for outcome 1
Time Frame: 10 minutes after lens insertion
Measure: Mean (Standard Deviation); unit: LogMAR units
Arm/Group | Lotrafilcon B | Senofilcon A | Omafilcon A | Balafilcon A
Number analyzed (Participants) | 35 | 35 | 35 | 35
LogMAR units | 0.14 (0.15) | 0.10 (0.15) | 0.15 (0.16) | 0.16 (0.19)
Statistical Analysis 1: Comparison: Lotrafilcon B vs Senofilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = 0.04, Standard Deviation 0.17
Statistical Analysis 2: Comparison: Lotrafilcon B vs Omafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.01, Standard Deviation 0.19
Statistical Analysis 3: Comparison: Lotrafilcon B vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.02, Standard Deviation 0.20
Statistical Analysis 4: Comparison: Senofilcon A vs Omafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.05, Standard Deviation 0.15
Statistical Analysis 5: Comparison: Senofilcon A vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.06, Standard Deviation 0.18
Statistical Analysis 6: Comparison: Omafilcon A vs Balafilcon A; Hypothesis is that visual acuity is the same for all lens types; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.05; p = 0.02, ANOVA; Mean Difference (Final Values) = -0.01, Standard Deviation 0.18

ADVERSE EVENTS:
Groups:
- Lotrafilcon B: lotrafilcon b toric contact lens
- Senofilcon A: senofilcon A toric contact lens
- Omafilcon A: omafilcon A toric contact lens
- Balafilcon A: balafilcon A toric contact lens
Arm/Group | Lotrafilcon B | Senofilcon A | Omafilcon A | Balafilcon A
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.